CLINICAL TRIAL: NCT05640193
Title: Pilot Trial of Lifileucel (LN-144) for Patients With Asymptomatic Melanoma Brain Metastases and Progression on Prior PD1 Therapy
Brief Title: A Study of LN-144 in People With Metastatic Melanoma to the Brain
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Iovance Biotherapeutics, Inc. (Industry); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-322
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Melanoma
Keywords: LN-144; Non-uveal melanoma; Lifileucel (LN-144); 22-322
MeSH Terms: conditions — Melanoma | interventions — lifileucel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Melanoma Brain Metastases (Experimental): Participants have melanoma brain metastases who will undergo surgical excision to generate LN-144.
  Interventions: Biological: Lifileucel (LN-144)

INTERVENTIONS:
Biological: Lifileucel (LN-144) — A portion of the patient's tumor is resected and serves as the starting material for manufacturing lifileucel. After preparative NMA-LD, patients are infused with their autologous TIL (lifileucel), followed by a short course of high-dose IL-2.

SUMMARY:
This is an open label study evaluating lifileucel (LN-144) in patients with melanoma brain metastases.

DETAILED DESCRIPTION:
Lifileucel (LN-144) is an autologous Tumor Infiltrating Lymphocytes (TIL) cell therapy that utilizes a 22-day centralized GMP process. Lifileucel is infused as part of a treatment regimen that includes preparative NMA-LD, followed by one-time autologous TIL infusion, and a short course of high-dose IL-2.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic melanoma with asymptomatic brain metastases
2. At least one resectable lesion (or aggregate of lesions resected) of a minimum 1.5 cm in diameter post-resection to generate TIL
3. Must be ≥ 18 years of age at time of consent
4. ECOG performance status of 0-1 and estimated life expectancy of ≥ 3 months
5. Adequate hematologic parameters and organ function

Exclusion Criteria:

1. Received organ allograft, except kidney transplant, or prior cell transfer therapy including TIL and CAR-T therapies
2. Ongoing grade 2-4 toxicity from prior immunotherapy (excluding endocrine, ocular toxicity or vitiligo)
3. History of hypersensitivity to any component or excipient of lifileucel or other treatment regimen drugs
4. Symptomatic brain metastases
5. Chronic systemic steroid therapy of > 10 mg/day
6. Active medical illness(es) that would pose increased risk for protocol participation
7. Must have negative syphilis assay and be seronegative for HIV, positive serology for HBV must have corresponding PCR assay and may be enrolled if viral load by PCR is undetectable
8. Primary immunodeficiency
9. Received live or attenuated vaccine within 28 days prior to beginning NMA-LD
10. Pregnant or breastfeeding
11. Patients who cannot receive gadolinium-enhanced MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Feasibility of treatment with LN-144 in patients with asymptomatic Metastatic Melanoma to the Brain (MMB) | 1 year
  measured by the number of patients who undergo surgery and successfully undergo LN-144 infusion

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Shoushtari, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm